CLINICAL TRIAL: NCT00566228
Title: Randomized, Double-Blind Phase III Clinical Trial Comparing Outcomes of Immunologic Autograft Engineering Versus Standard Autograft Collection in Patients Undergoing Autologous Stem Cell Transplantation for Lymphoma
Brief Title: Two Different Methods of Collecting Stem Cells For an Autologous Stem Cell Transplant in Treating Patients With Diffuse Large Cell Lymphoma
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Mayo Clinic (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: MC0681; P30CA015083 (NIH); MC0681 (Other: Mayo Clinic Cancer Center); 07-000789 (Other: Mayo Clinic IRB)
Record Dates: First submitted 2007-11-30; First posted 2007-12-03 (Estimated); Results first posted 2018-07-09 (Actual); Last update posted 2018-07-09 (Actual); Status verified 2018-06

CONDITIONS: Lymphoma
Keywords: noncontiguous stage II adult diffuse large cell lymphoma; stage III adult diffuse large cell lymphoma; stage IV adult diffuse large cell lymphoma; recurrent adult diffuse large cell lymphoma
MeSH Terms: conditions — Lymphoma; Lymphoma, Large B-Cell, Diffuse | interventions — Leukapheresis

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Immunologic autograft engineering (Experimental): Patients' stem cells are collected according to modified Amicus settings (i.e., MNC OFFSET = 0.0 and RBC = 7.0). Patients undergo ASCT IV on the day of apheresis (lymphocyte enriched autograft).
  Interventions: Procedure: autologous hematopoietic stem cell transplantation; Procedure: leukapheresis
- Standard autograft collection (Active Comparator): Patients' stem cells are collected according to standard Amicus settings (i.e., MNC OFFSET = 1.5 and RBC OFFSET = 5.0). Patients undergo ASCT IV on the day of apheresis.
  Interventions: Procedure: autologous hematopoietic stem cell transplantation; Procedure: leukapheresis

INTERVENTIONS:
Procedure: autologous hematopoietic stem cell transplantation — Patients undergo autologous stem cell transplantation
Procedure: leukapheresis — Stem cells collected

SUMMARY:
RATIONALE: It is not yet known which method of stem cell collection is best for patients undergoing an autologous stem cell transplant.

PURPOSE: This randomized phase III trial is comparing two different methods of collecting stem cells in patients undergoing stem cell transplant for diffuse large cell lymphoma.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* Determine the therapeutic effect of instrument-driven lymphocyte enrichment of the autograft absolute lymphocyte count (A-ALC) compared to "standard autograft collection" as determined by progression-free survival post-transplantation.

Secondary

* Determine the profile of immune effector cells of the "lymphocyte enriched autograft" vs "standard autograft" and peripheral blood after autologous stem cell transplant (ASCT) and their impact on post- ASCT immunological reconstitution and clinical endpoints.
* Perform quantitative and functional analysis of T, B, NK, and dendritic cells from the apheresis product and peripheral blood samples at multiple timepoints after transplantation.
* Determine and compare the proportion of patients who are progression-free and alive at 1 and 2 years.
* Determine the differences in overall survival between the two collection method arms.
* Evaluate and characterize differences in transplantation outcomes (e.g., time to ALC engraftment, incidence of infection, and the CD34 count) between the two collection method arms.

OUTLINE: Patients are stratified according to baseline International Prognostic Factor (≥ 2 factors vs < 2 factors) and PET scan findings prior to transplantation (positive vs negative). Patients receive filgrastim (G-CSF) alone or G-CSF and sargramostim (GM-CSF) daily for stem cell mobilization. Once the peripheral CD34-positive cell count reaches ≥ 10/μL, patients undergo stem cell collection. Patients are then randomized to 1 of 2 treatment arms for standard autologous stem cell transplantation (ASCT).

* Immunologic autograft engineering: Patients' stem cells are collected according to modified Amicus settings (i.e., MNC OFFSET = 0.0 and RBC = 7.0). Patients undergo ASCT IV on the day of apheresis (lymphocyte enriched autograft).
* Standard autograft collection: Patients' stem cells are collected according to standard Amicus settings (i.e., MNC OFFSET = 1.5 and RBC OFFSET = 5.0). Patients undergo ASCT IV on the day of apheresis.

Patients undergo blood sample collection periodically for immunological studies. Samples are analyzed for immunophenotyping of immune cell subsets via multicolor flow cytometry, immunoglobulin reconstitution, and functional T-cell immunity.

After completion of study treatment, patients are followed at day 15 post ASCT and then at 3, 6, 9, and 12 months.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Diagnosis of diffuse large cell lymphoma

  * Low-grade non-Hodgkin lymphoma transformed to diffuse large cell lymphoma allowed
* Candidate for with autologous peripheral blood stem cell transplantation

  * Not requiring bone marrow harvest to collect stem cells
  * No chemotherapy with filgrastim ( G-CSF) or mobilization study drug (i.e., AMD3100) needed for mobilization of stem cells

PATIENT CHARACTERISTICS:

* ECOG performance status 0-1
* Cardiac and pulmonary status sufficient to undergo apheresis and stem cell transplantation
* Negative pregnancy test
* Not pregnant or nursing
* Fertile patients must use effective contraception
* HIV negative
* No active uncontrolled infection requiring antibiotic treatment
* No comorbid condition which, in view of the investigators, renders the patient at high risk from treatment complications
* Willing to provide all research blood samples as required by the protocol

PRIOR CONCURRENT THERAPY:

* At least 4 weeks since prior chemotherapy (rituxan is not considered chemotherapy for the purpose of this study)
* More than 4 weeks since prior experimental therapy
* No concurrent enrollment on another experimental protocol during the mobilization phase
* No concurrent participation in any autologous stem cell transplantation study that is not using the standard conditioning regimens for lymphomas

Ages: 18 Years to 120 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 122 (Actual)
Dates: Start 2007-12; Primary Completion 2015-01-15 (Actual); Study Completion 2015-01-15 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Luis F. Porrata, MD, Study Chair — Mayo Clinic
Locations (1):
- Mayo Clinic, Rochester, Minnesota, United States

REFERENCES:
- [Result] Porrata LF, Burgstaler EA, Winters JL, Jacob EK, Gastineau DA, Suman VJ, Inwards DJ, Ansell SM, Micallef IN, Johnston PB, Nevala W, Markovic SN. Immunologic Autograft Engineering and Survival in Non-Hodgkin Lymphoma. Biol Blood Marrow Transplant. 2016 Jun;22(6):1017-1023. doi: 10.1016/j.bbmt.2016.01.024. Epub 2016 Jan 27. PMID 26826432
- [Derived] Porrata LF, Inwards DJ, Ansell SM, Micallef IN, Johnston PB, Villasboas JC, Markovic SN. Autograft immune content and survival in non-Hodgkin's lymphoma: A post hoc analysis. Leuk Res. 2019 Jun;81:1-9. doi: 10.1016/j.leukres.2019.03.009. Epub 2019 Apr 4. PMID 30978434

RESULTS

PARTICIPANT FLOW:
Groups:
- Immunologic Autograft Engineering: Patients' stem cells are collected according to modified Amicus settings (i.e., MNC OFFSET = 0.0 and RBC = 7.0).
- Standard Autograft Collection: Patients' stem cells are collected according to standard Amicus settings (i.e., MNC OFFSET = 1.5 and RBC OFFSET = 5.0).
Period: Overall Study
Arm/Group | Immunologic Autograft Engineering | Standard Autograft Collection
Started | 62 | 60
Completed | 56 | 55
Not Completed | 6 | 5
Not completed — Withdrawal by Subject | 1 | 0
Not completed — Attempt to mobilize stem cells failed | 2 | 2
Not completed — Unable to collect sufficient CD34 cells | 3 | 2
Not completed — progressed before infusion could occur | 0 | 1

BASELINE CHARACTERISTICS:
Population: All patients who started the study and did not withdraw consent prior to the start of treatment were included.
Groups:
- Total: Total of all reporting groups
Arm/Group | Immunologic Autograft Engineering | Standard Autograft Collection | Total
Number analyzed (Participants) | 61 | 60 | 121
Age, Continuous [Median (Inter-Quartile Range); unit: years] | 58 [50 to 64] | 58 [49 to 64] | 58 [50 to 64]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 16 | 20 | 36
  Male | 45 | 40 | 85
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 61 | 60 | 121

OUTCOME MEASURES:

1. Primary Outcome: Median Progression-free Survival
Description: Progression free survival (PFS) was defined as the time from the date of infusion to disease progression, relapse, or death from any cause. Patients alive without disease progression or relapse were censored at their last disease evaluation or at their secondary primary cancer diagnosis, whichever occurred first. Criteria for Relapsed Disease: Appearance of any new lesion or increase by ≥50% in the size of previously involved sites, ≥50% increase in greatest diameter of any previously identified node >1.0 cm in its short axis or in the sum of the products of diameters (SPD) of more than one node. Criteria for Progressive Disease: ≥50% increase from nadir in the SPD of any previously identified abnormal node or ALC for partial remissions or non-responders, Appearance of any new lesion (≥ 2x2 cm). A log rank test was used to assess whether PFS differed with respect to apheresis collection method.
Time Frame: Date of infusion to disease progression, relapse, or death from any cause whichever came first, assessed up to 24 months post enrollment.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Immunologic Autograft Engineering | Standard Autograft Collection
Number analyzed (Participants) | 56 | 55
months | NA [NA to NA] — The median and 95% confidence interval was not reached. | NA [NA to NA] — The median and 95% confidence interval was not reached.
Statistical Analysis 1: Comparison: Immunologic Autograft Engineering vs Standard Autograft Collection; Test type: Superiority; p = 0.690, Log Rank; Hazard Ratio (HR) = 1.13, 95% CI 2-sided [0.62 to 2.08]

2. Secondary Outcome: Progression-free Survival Rate at 1 Year
Description: Progression-free survival rate (percentage) at one year is defined as 100 times the number of patients who have not progressed, relapsed and/or died divided by the total number of evaluable patients in each arm. Criteria for Relapsed Disease: Appearance of any new lesion or increase by ≥50% in the size of previously involved sites, ≥50% increase in greatest diameter of any previously identified node >1.0 cm in its short axis or in the SPD of more than one node. Criteria for Progressive Disease: ≥50% increase from nadir in the SPD of any previously identified abnormal node or ALC for partial remissions or non-responders, Appearance of any new lesion (≥ 2x2 cm).
Time Frame: Date of infusion to disease progression, relapse, or death from any cause, up to one year
Measure: Number (95% Confidence Interval); unit: percentage of patients
Arm/Group | Immunologic Autograft Engineering | Standard Autograft Collection
Number analyzed (Participants) | 56 | 55
percentage of patients | 73.1 [62.3 to 85.7] | 65.4 [53.9 to 79.3]

3. Secondary Outcome: Progression-free Survival Rate at 2 Years
Description: Progression-free survival rate (percentage) at two years is defined as 100 times the number of patients who have not progressed, relapsed and/or died divided by the total number of evaluable patients in each arm. Criteria for Relapsed Disease: Appearance of any new lesion or increase by ≥50% in the size of previously involved sites, ≥50% increase in greatest diameter of any previously identified node >1.0 cm in its short axis or in the SPD of more than one node. Criteria for Progressive Disease: ≥50% increase from nadir in the SPD of any previously identified abnormal node or ALC for partial remissions or non-responders, Appearance of any new lesion (≥ 2x2 cm).
Time Frame: Date of infusion to disease progression, relapse, or death from any cause, up to two years
Measure: Number (95% Confidence Interval); unit: percentage of patients
Arm/Group | Immunologic Autograft Engineering | Standard Autograft Collection
Number analyzed (Participants) | 56 | 55
percentage of patients | 57.9 [46.1 to 72.7] | 65.4 [53.9 to 79.3]

4. Secondary Outcome: One-year Overall Survival Rate
Description: Overall survival (OS) was defined at the time from infusion to death from any cause. The one-year OS rate is defined as the percentage of patients who are still alive after one year. A log rank test was used to assess whether OS differed with respect to apheresis collection method.
Time Frame: date of infusion to death from any cause, up to one year
Measure: Number (95% Confidence Interval); unit: percentage of patients
Arm/Group | Immunologic Autograft Engineering | Standard Autograft Collection
Number analyzed (Participants) | 56 | 55
percentage of patients | 91.1 [83.9 to 98.9] | 83.6 [74.4 to 94.0]
Statistical Analysis 1: Comparison: Immunologic Autograft Engineering vs Standard Autograft Collection; Test type: Superiority; p = 0.679, Log Rank

5. Secondary Outcome: Median Time to Absolute Lymphocyte Count Engraftment
Description: The time to absolute lymphocyte count (ALC) engraftment will be evaluated and compared between the two arms, where time to ALC engraftment is defined as the time from transplant to the time they achieve ALC > 500.
Time Frame: Up to 30 days after autologous peripheral hematopoietic stem cell transplantation
Measure: Median (Full Range); unit: days
Arm/Group | Immunologic Autograft Engineering | Standard Autograft Collection
Number analyzed (Participants) | 56 | 55
days | 14 [10 to 30] | 14 [10 to 30]

6. Secondary Outcome: Median Number of CD34 Cells/kg Infused
Description: Five (5) to seven (7) days after patient received granulocyte-colony stimulating factor and reached a peripheral CD34 count of 10 cells/microliter or greater, stem cell collection began. Apheresis collections were to be performed daily. At least 2 x 10^6 CD34 cells/kg were to be collected. Additional collections were at the discretion of the transplantation team. The median number of CD34 cells/kg infused are reported for each arm below.
Time Frame: 5 to 7 days after patient received granulocyte-colony stimulating factor and reached a peripheral CD34 count of 10 cells/microliter or greater
Measure: Median (Full Range); unit: x10^6 cells/kg
Arm/Group | Immunologic Autograft Engineering | Standard Autograft Collection
Number analyzed (Participants) | 56 | 55
x10^6 cells/kg | 4.6 [2.0 to 8.2] | 5.3 [3.0 to 11.4]

7. Other Pre Specified Outcome: Evaluation and Comparison of Immunologic Recovery Within and Between the Arms by Assessing the Quantitative and Functional Immune Effector Cells (T, B, or NK Cells) From the Apheresis Product
Description: Evaluation and comparison of immunologic recovery within and between the arms by assessing the quantitative and functional immune effector cells (T, B, or NK cells) from the apheresis product
Time Frame: Baseline
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: At completion of apheresis collection; Up to 2 years.
Description: CTCAE term (AE description) and grade: The descriptions and grading scales found in the revised NCI Common Terminology Criteria for Adverse Events (CTCAE) version 3.0 will be utilized for AE reporting. Each CTCAE term in the current version is a unique representation of a specific event used for medical documentation and scientific analysis and is a single MedDRA Lowest Level Term (LLT).
Arm/Group | Immunologic Autograft Engineering | Standard Autograft Collection
All-Cause Mortality (participants affected / at risk) | 0/57 | 0/57
Serious Adverse Events (participants affected / at risk) | 0/57 | 0/57
Other Adverse Events (participants affected / at risk) | 22/57 | 17/57
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Immunologic Autograft Engineering (N=57) | Standard Autograft Collection (N=57)
Hemoglobin decreased (Blood and lymphatic system disorders) | 5 (5) | 4 (4)
Atrial fibrillation (Cardiac disorders) | 1 (1) | 0 (0)
Atrial tachycardia (Cardiac disorders) | 1 (1) | 0 (0)
Injection site reaction (General disorders) | 0 (0) | 3 (3)
Bruising (Injury, poisoning and procedural complications) | 11 (11) | 9 (9)
Platelet count decreased (Investigations) | 6 (6) | 4 (4)
Peripheral sensory neuropathy (Nervous system disorders) | 5 (5) | 6 (6)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes